CLINICAL TRIAL: NCT06265558
Title: Prevention of Postoperative Complications by Negative Pressure Therapy After Complex Breast Cancer Surgery: a Prospective Randomized Controlled Trial
Brief Title: Prevention of Postoperative Complications by Negative Pressure Therapy After Complex Breast Cancer Surgery
Acronym: TPN-SEIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2023-08 TPN
Record Dates: First submitted 2024-02-07; First posted 2024-02-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Pressure negative therapy; Breast surgery; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Negative-Pressure Wound Therapy; Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Conventional post-operative care
  Interventions: Procedure: Dressing
- Negative pressure therapy (NPT) (Experimental): Immediate post-operative negative pressure therapy
  Interventions: Procedure: Negative pressure therapy (NPT)

INTERVENTIONS:
Procedure: Negative pressure therapy (NPT) — Negative pressure therapy (NPT) involves placing the surface of a wound under a pressure lower than the ambient atmospheric pressure. To achieve this, a specially designed dressing is connected to a vacuum source and an exudate collection system.
  Arms: Negative pressure therapy (NPT)
Procedure: Dressing — Fatty dressing or hydrocellular dressing
  Arms: Standard care

SUMMARY:
There is little scientific data concerning the use of negative pressure therapy after immediate breast reconstruction.

That strategy of treatment-reconstruction has expanded increasingly since the last years.

The current literature reports only 3 studies on the use of preventive negative pressure therapy in oncologic breast surgery.

Moreover, all three are retrospective, case-control studies with serious limitations.

The largest published series reports a reduction in the overall complication rate from 15.9% to 8.5%, and a significant reduction in several criteria: infection, scar dehiscence and necrosis. However, the study presents significant biases, with non-comparable populations in terms of comorbidities, surgical procedure performed, inclusion periods (and therefore experience in performing oncological surgery).

There was also a high probability of under-assessment or postponement of post-operative complications, which is typical of published retrospective surgical studies.

The published results therefore strongly encourage further investigation of negative pressure therapy in oncological breast surgery.

DETAILED DESCRIPTION:
In 2022, excisional surgery is still one of the mainstays of breast cancer treatment. The excisional surgery is often combined with adjuvant treatments, which may include medical treatments such as chemotherapy, targeted therapies and immunotherapy, hormone therapy and radiotherapy. All these treatments have toxicities that impact on patients' quality of life.

One of the main complications of surgery is scarring. The rate is around 2% for "simple" breast surgery (conservative breast surgery - total mastectomy). This rate can rise sharply in the case of "complex" breast surgery, such as high-level oncoplasty, or mastectomy with Immediate Breast Reconstruction (IBR). This rate of surgical wound complications (ischemia, necrosis, dehiscence, infection) reached 20% in our local series of Immediate Breast Reconstruction (IBR) by prosthesis. This rate may exceed 30% in some series, depending on the surgical technique and the population, in cases of smoking, diabetes, previous radiotherapy, obesity and large breast volume. The increasing prevalence of these risk factors in the population means that scarring disorders must be taken into account in daily cancer care.

The impact of these scarring disorders is manifold:

* Delayed initiation of adjuvant therapy with an impact on overall survival.
* Cosmetic impact of scarring
* Possible loss of prosthetic breast reconstruction
* Patient dissatisfaction, with increased burden of care
* Overall impact on patient quality of life
* Economic impact linked to the length of care over time (consumption of dressing materials and personal time) Preventing the onset of wound-healing disorders is therefore vital in order to avoid these multiple consequences for the patient and the healthcare system.

In breast surgery, the use of preventive NPT (Negative Pressure Therapy) has been little studied. The NPT has been used mainly in cosmetic surgery procedures such as breast reduction, with results in favor of NPT. The most comprehensive study is a multicenter randomized trial which included 200 patients scheduled for bilateral breast reduction. In this trial, the comparison was made between the 2 breasts, each patient being her own control. The calculation of the number of subjects was based on a reduction in the complication rate from 20% to 10% (i.e., a 50% reduction). The study was positive, showing a reduction in the dehiscence rate at day 21 from 26% to 16%. In this study, patients were under-selected, and around 40% had risk factors for complications. A second randomized study, with similar methodology and judgment criteria, included 32 patients undergoing bilateral breast reduction. The results of this study are significant, but unfortunately there weren't much detail in the publication.

There is little scientific data concerning the use of negative pressure therapy after immediate breast reconstruction. There are very few data on the use of Negative pressure Therapy (NPT) after immediate Breast Reconstruction (IBR), a treatment-reconstruction strategy that has been expanding rapidly since recent years. The current literature reports only 3 studies on the use of preventive Negative pressure Therapy (NPT) in oncologic breast surgery. All three are retrospective, case-control studies with serious limitations. The largest published series involved 356 patients and 665 breasts. A reduction was reported in the overall complication rate from 15.9% to 8.5%, and a significant reduction in several criteria: infection, seroma, scar dehiscence and necrosis. However, the study presents significant biases, with non-comparable populations in terms of co-morbidities, surgical procedure performed, inclusion periods (and therefore experience in performing oncological surgery). There was also a high probability of under-assessment or postponement of post-operative complications, which is typical of published retrospective surgical studies.

The published results therefore strongly encourage further investigation of Negative Pressure Therapy (NPT) in oncological breast surgery.

Our hypothesis, then, is that preventive NPT in the immediate post-operative phase of complex breast surgery can prevent the onset of post-operative scarring disorders and shorten the time to complete healing.

To date, there are no randomized prospective studies of NPT in complex oncologic breast surgery. Randomized studies already published in general surgery provide a good level of evidence for the efficacy of NPT in preventing local post-operative complications. The latest systematic review and meta-analysis found a reduction in the risk of surgical site infection, from 13% to 8.8%, all types of surgery included. The benefit on the risk of dehiscence in general surgery is less strong, but a 30% reduction was found in a meta-analysis of studies involving only a preventive NPT device, a device widely used throughout the world.

In view of these results from randomized trials in general surgery and non-oncological breast surgery, and the results of retrospective studies in oncological breast surgery, a randomized trial must be carried out. This randomized controlled trial will be pragmatic, incorporating an intermediate analysis, given the endpoint evaluating the reduction in complications in a surgical context, to rapidly meet our objectives with a sufficient level of evidence to have an immediate impact on patients and modify practice.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 years
2. Patient with unilateral invasive or in situ breast carcinoma
3. Patient with or without neoadjuvant treatment
4. Patient presenting an indication for complex breast surgery by mastectomy with immediate breast reconstruction by implant or oncoplasty by T-shaped mammoplasty.
5. Patient presenting at least one of the following risk factors for scarring disorders:

   * Obesity with Body Mass Index BMI ≥ 30 and/or Cup size ≥ E
   * Active smoking or smoking cessation for less than one month
   * Diabetes
   * History of homolateral breast radiotherapy
   * Long-term corticosteroid therapy
6. Patient to have signed informed consent prior to study entry
7. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
8. Patient affiliated with a health insurance plan.

Exclusion Criteria:

1. Legal incapacity or limited legal capacity. Medical or psychological conditions preventing the patient from completing the study or signing the consent form.
2. Pregnant or breast-feeding patient as determined in medical records as part of standard patients care and follow-up
3. Patient under guardianship or safeguard of justice
4. Patient participating in an interventional study with the objective of wound healing
5. Any concurrent or planned surgical procedure on the contralateral breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 254 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rate of patients experiencing postoperative wound healing complication | From baseline to 30 days after surgery
  defined as the presence of at least one of the following criteria: Deep postoperative infection of the prosthetic pocket (confirmed by a positive bacterial culture with a pathogen commonly associated with surgical site infections), wound dehiscence, or incomplete wound healing at postoperative day 30 (D30). The primary endpoint is a composite criterion (dehiscence, infection, or delayed wound healing at D30), with negative pressure wound therapy expected to reduce each complication individually. This composite endpoint capture overall postoperative wound healing complications by integrating multiple clinically relevant events into a single measure.

SECONDARY OUTCOMES:
Rate of patients with a surgical site infection | From baseline to 90 days after the surgery
  Number of patients with surgical site infection divided by total number of patients operated on in the trial.
Surgical revision rate | From baseline to 90 days after the surgery
  Number of patients with repeat surgery divided by the total number of patients operated on in the trial.
Incidence of patients with at least one hospital readmission | Frm baseline to 90 days after the surgery
  Number of patients with at least one hospital readmission divided by total number of patients operated on in the trial.
Surgical complication rate according to the National Cancer Institute - Common Terminology Criteria for Adverse Events version 5 classification | Approximately 10 days, from surgery to hospital discharge
  The NCI CTC classification is used for grading adverse events which occur as a result of trial procedures. It includes 5 grades from grade 1 (recourse to usual postoperative treatments) to Grade 5 (death).
Time to initiation of adjuvant therapy | Approximately 3 months, from surgery to beginning of adjuvant therapy
  Number of days between surgery and initiation of adjuvant therapy
Quality of life evaluated by questionnaire QLQ-C30 (Version 3) | From baseline to 15 days then to 30 and 90 days after surgery
  The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients.Version 3, incorporates five functional scales on physical (PF), role (RF), cognitive (CF), emotional (EF) and social (SF) functioning, three symptom scales on fatigue (FA), pain (PA) and nausea and vomiting (NV), single items assessing dyspnoea (DY), insomnia (SL), loss of appetite (AP), constipation (CO) and diarrhoea (DI), one item assessing perceived financial impact (FI) and a global health status/QoL scale (Global QoL). Each item is scored in one of four categories 1) 'Not at all', 2) 'A little', 3) 'Quite a bit' 4) 'Very much', with the exception of 'Global QoL'which ranges from 1) 'Very poor' to 7) 'Excellent'.
  Scoring of the items in the PF scale in the latest revision of EORTC QLQ-C30, Version 3 is extended to the four-point scale instead of the previous 'Yes/No' dichotomy
Quality of life evaluated by questionnaire QLQ-BReast cancer (BR23) | From baseline to 15 days then to 30 and 90 days after surgery
  The Breast Cancer module is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-BR23 incorporates five multi-item scales to assess body image, sexual functioning, systemic therapy side effects, breast symptoms, and arm symptoms. All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, whilst a high score for the symptom scales represents a high level of symptomatology or problems.
Patient satisfaction with cosmetic result evaluated using the BR23 questionnaire | From baseline to 15 days then to 30 and 90 days after surgery
  The QLQ-BR23 incorporates five multi-item scales to assess body image, sexual functioning, systemic therapy side effects, breast symptoms, and arm symptoms.
Medical cost of post-surgery care | From baseline to 90 days after surgery
  A comparison will be conducted between the two study arms. The cost of post-operative care will be calculated based on data including the number and type of dressings, consumables, nursing time, reasons for hospital consultations and hospitalisations, and mode of transport in relation to the distance between the patient's home and the hospital
Time to complete wound healing | From surgery to 30 days post-surgery
  It will be evaluated clinically by surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Mathias NERON, MD, Study Chair — Institut régional du Cancer de Montpellier (ICM)
Locations (7):
- France (7):
  - Centre Georges-François Leclerc, Dijon, Côte d'Or
  - Centre Hospitalier de Nîmes, Nîmes, GARD
  - Institut Bergonié, Bordeaux, Gironde
  - Centre Hospitalier de Montpellier, Montpellier, Hérault
  - Institut régional du Cancer de Montpellier, Montpellier, Hérault
  - Institut de Cancérologie de l'Ouest, Angers, Maine Et Loire
  - Centre Léon Bérard, Lyon, Rhône

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be made available on request and with the completion of a contract between the sponsor and the requester.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Access to study data upon written detailed request sent to the institute of Montpellier Cancer (ICM), following publication and until 5 years after publication of summary data.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Bowen ME, Mone MC, Buys SS, Sheng X, Nelson EW. Surgical Outcomes for Mastectomy Patients Receiving Neoadjuvant Chemotherapy: A Propensity-Matched Analysis. Ann Surg. 2017 Mar;265(3):448-456. doi: 10.1097/SLA.0000000000001804. PMID 27280515
- [Background] Clough KB, Kaufman GJ, Nos C, Buccimazza I, Sarfati IM. Improving breast cancer surgery: a classification and quadrant per quadrant atlas for oncoplastic surgery. Ann Surg Oncol. 2010 May;17(5):1375-91. doi: 10.1245/s10434-009-0792-y. Epub 2010 Feb 6. PMID 20140531
- [Background] Donovan CA, Harit AP, Chung A, Bao J, Giuliano AE, Amersi F. Oncological and Surgical Outcomes After Nipple-Sparing Mastectomy: Do Incisions Matter? Ann Surg Oncol. 2016 Oct;23(10):3226-31. doi: 10.1245/s10434-016-5323-z. Epub 2016 Jun 28. PMID 27352202
- [Background] Bleicher RJ, Moran MS, Ruth K, Edge SB, Dietz JM, Wilke LG, Stearns V, Kurtzman SH, Klein J, Yao KA. The Impact of Radiotherapy Delay in Breast Conservation Patients Not Receiving Chemotherapy and the Rationale for Dichotomizing the Radiation Oncology Time-Dependent Standard into Two Quality Measures. Ann Surg Oncol. 2022 Jan;29(1):469-481. doi: 10.1245/s10434-021-10512-1. Epub 2021 Jul 29. PMID 34324114
- [Background] Gagliato Dde M, Gonzalez-Angulo AM, Lei X, Theriault RL, Giordano SH, Valero V, Hortobagyi GN, Chavez-Macgregor M. Clinical impact of delaying initiation of adjuvant chemotherapy in patients with breast cancer. J Clin Oncol. 2014 Mar 10;32(8):735-44. doi: 10.1200/JCO.2013.49.7693. Epub 2014 Jan 27. PMID 24470007
- [Background] Galiano RD, Hudson D, Shin J, van der Hulst R, Tanaydin V, Djohan R, Duteille F, Cockwill J, Megginson S, Huddleston E. Incisional Negative Pressure Wound Therapy for Prevention of Wound Healing Complications Following Reduction Mammaplasty. Plast Reconstr Surg Glob Open. 2018 Jan 12;6(1):e1560. doi: 10.1097/GOX.0000000000001560. eCollection 2018 Jan. PMID 29464150
- [Background] Tanaydin V, Beugels J, Andriessen A, Sawor JH, van der Hulst RRWJ. Randomized Controlled Study Comparing Disposable Negative-Pressure Wound Therapy with Standard Care in Bilateral Breast Reduction Mammoplasty Evaluating Surgical Site Complications and Scar Quality. Aesthetic Plast Surg. 2018 Aug;42(4):927-935. doi: 10.1007/s00266-018-1095-0. Epub 2018 Feb 13. PMID 29442143
- [Background] Johnson ON 3rd, Reitz CL, Thai K. Closed Incisional Negative Pressure Therapy Significantly Reduces Early Wound Dehiscence after Reduction Mammaplasty. Plast Reconstr Surg Glob Open. 2021 Mar 22;9(3):e3496. doi: 10.1097/GOX.0000000000003496. eCollection 2021 Mar. PMID 33968556
- [Background] Cagney D, Simmons L, O'Leary DP, Corrigan M, Kelly L, O'Sullivan MJ, Liew A, Redmond HP. The Efficacy of Prophylactic Negative Pressure Wound Therapy for Closed Incisions in Breast Surgery: A Systematic Review and Meta-Analysis. World J Surg. 2020 May;44(5):1526-1537. doi: 10.1007/s00268-019-05335-x. PMID 31900568
- [Background] Chicco M, Huang TC, Cheng HT. Negative-Pressure Wound Therapy in the Prevention and Management of Complications From Prosthetic Breast Reconstruction: A Systematic Review and Meta-analysis. Ann Plast Surg. 2021 Oct 1;87(4):478-483. doi: 10.1097/SAP.0000000000002722. PMID 34060773
- [Background] Gabriel A, Sigalove S, Sigalove N, Storm-Dickerson T, Rice J, Maxwell P, Griffin L. The Impact of Closed Incision Negative Pressure Therapy on Postoperative Breast Reconstruction Outcomes. Plast Reconstr Surg Glob Open. 2018 Aug 7;6(8):e1880. doi: 10.1097/GOX.0000000000001880. eCollection 2018 Aug. PMID 30324063
- [Background] Norman G, Goh EL, Dumville JC, Shi C, Liu Z, Chiverton L, Stankiewicz M, Reid A. Negative pressure wound therapy for surgical wounds healing by primary closure. Cochrane Database Syst Rev. 2020 Jun 15;6(6):CD009261. doi: 10.1002/14651858.CD009261.pub6. PMID 32542647
- [Background] Saunders C, Nherera LM, Horner A, Trueman P. Single-use negative-pressure wound therapy versus conventional dressings for closed surgical incisions: systematic literature review and meta-analysis. BJS Open. 2021 Jan 8;5(1):zraa003. doi: 10.1093/bjsopen/zraa003. PMID 33609382
- [Background] Neron M, Delmond L, Gourgou S, Delaine S, Chalbos P, Moussion A, Taoum C. Prevention of postoperative complications with negative pressure wound therapy after complex breast cancer surgery: a study protocol of a randomised controlled trial (TPN-SEIN). BMJ Open. 2026 Jan 3;16(1):e103827. doi: 10.1136/bmjopen-2025-103827. PMID 41485781
- See also: Breast cancers - Recommendations and practice aids — https://www.e-cancer.fr/Professionnels-de-sante/Recommandations-et-outils-d-aide-a-la-pratique/Cancers-du-sein
- See also: French Society of Senology and Breast Pathology multimedia library — http://medias.sfspm.org/Lyon-2021/Programme/2/Enseignements-en-Chirurgie/